CLINICAL TRIAL: NCT00591331
Title: Phase 1 Evaluation of the Phototoxic Potential of NatrOVA Creme Rinse - 1% in Healthy Volunteers
Brief Title: Phototoxicity Potential of NatrOVA Creme Rinse - 1%
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Responsible Party: David C. Rowe, ParaPRO, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPN-107-07; HTR 07-128384-111
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2007-12

CONDITIONS: Head Lice
Keywords: Head Lice
MeSH Terms: interventions — spinosad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): NatrOVA Creme Rinse - 1%
  Interventions: Drug: Spinosad (the active ingredient in NatrOVA)
- 2 (Experimental): NatrOVA Creme Rinse Vehicle Only
  Interventions: Drug: Spinosad (the active ingredient in NatrOVA)
- 3 (Placebo Comparator): Blank patch
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Spinosad (the active ingredient in NatrOVA) — This is a patch test in which the test material is applied to the patch and the patch applied to the skin.
  Arms: 1; 2
Drug: placebo
  Arms: 3

SUMMARY:
This study will evaluate the primary irritation potential of NatrOVA Creme Rinse - 1% in humans, after exposure to UV radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18-65 years of age and in good health.
2. Fitzpatrick skin type I, II or III

Exclusion Criteria:

1. History of severe reactions from exposure to sunlight
2. Known allergies or sensitivities to adhesives in patches
3. Inability to evaluate the skin in and around the test sites
4. Diabetes requiring medication
5. Clinical significant skin disease
6. Asthma or other severe respiratory disease
7. Known immunological disorders such as HIV, AIDS, lupus,rheumatoid arthritis
8. History or current skin cancer
9. Mastectomy for cancer involving removal of lymph nodes draining the test sites
10. Epilepsy
11. Pregnancy, lactation, or planned pregnancy during study period
12. Chronic use of systemic antihistamine medication within 14 days of screening
13. Use of anti-inflammatory drugs within 2 days of Screening Visit 1
14. Currently receiving allergy injections
15. Use of immunosuppressive drugs
16. Topical drugs used at the test site within 7 days of Screening Visit 1
17. Current participation in any clinical trial
18. Participation in any patch test for irritation or sensitization or UV exposures within 4 weeks of study start
19. Use of any investigational drug therapy within 4 weeks of study start.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety endpoint will be visual grading of UV irradiated test sites and assessments of adverse experiences | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: John V Murray, MD, Principal Investigator — Hill Top Research
Locations (1):
- Hill Top Research, St. Petersburg, Florida, United States

REFERENCES:
- See also: sponsor web site — http://www.parapro.com